CLINICAL TRIAL: NCT00276289
Title: Spironolactone to Decrease Potassium Wasting in Hypercalciuric Patients Treated With Thiazide Diuretics
Brief Title: Spironolactone to Decrease Potassium Wasting in Hypercalciurics on Thiazides Diuretics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0509-05
Record Dates: First submitted 2006-01-11; First posted 2006-01-13 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2009-12

CONDITIONS: Idiopathic Hypercalciuria; Hypokalemia Caused by Thiazide Diuretics
Keywords: nephrolithiasis; hypercalciuria; hypokalemia; thiazide diuretics
MeSH Terms: conditions — Nephrolithiasis; Hypercalciuria; Hypokalemia | interventions — Spironolactone

INTERVENTIONS:
Drug: Spironolactone

SUMMARY:
Kidney stone formation due to an excess of calcium in the urine is a common problem. It is treated with thiazide diuretics. These drugs often cause excessively low blood potassium levels that in turn require large doses of potassium supplements. These supplements are often large, unpleasant and easy to forget. We are trying the addition of spironolactone to these patients' medications to see if it allows them to take a lower dose of potassium.

DETAILED DESCRIPTION:
See rationale above

Ten patients who have had multiple kidney stones primarily due to hypercalciuria and who are currently on stable dose of thiazide or thiazide plus amiloride will be enrolled in the study. In addition, pts have to require at least 60mEq of K supplementation a day or be on 40mEq and be hypokalemic and unable to tolerate increased K supplements. We will then give them 50mg a day of spironolactone for four weeks. A complete 24-hour urine stone profile will be obtained before and after the drug is administered. After four weeks the patients' serum potassium will be rechecked, and their dose will be lowered according to a nomogram.

Primary end point is the mean change in serum K before and after spironolactone. Secondary endpoints are the change in urine calcium on and off the drug and the mean reduction in K dose on the drug.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* History of idiopathic hypercalciuria (>200mg per 24 hours or a Ca/cr ratio of >140) felt to be the primary etiology of patient's kidney stones
* History of at least three kidney stone events
* On same dose of thiazide diuretic for at least three months
* On stable dose of K 60mEq or more a day to maintain serum K >3.5 or unable to tolerate an increase in K supplement with dose at least 40mEq a day

Exclusion Criteria:

* Use of ACE inhibitor, ACE receptor blocker or other medication known to effect serum potassium levels
* GFR <80 by MDRD equation
* Serious cardiac disease, diabetes, CKD , current or planned pregnancy or breastfeeding
* History of hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-01; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Change in serum potassium on spironolactone versus off of it

SECONDARY OUTCOMES:
change in urinary calcium excretion
mean reduction in dose of potassium supplements

CONTACTS AND LOCATIONS:
Overall Officials: Sharon S Moe, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Department of Medicine, Division of Nephrology, Indianapolis, Indiana, United States